CLINICAL TRIAL: NCT02924779
Title: An Observational Study Investigating the Influence of Physical Position of Epidural Catheters and Their Function During Labour Analgesia
Brief Title: An Observational Study Investigating the Positioning of Epidural Catheters and Their Function During Labour Analgesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rotkreuzklinikum München gGmbH (Other)
Responsible Party: Principal Investigator, Ellis Muggleton, Anaesthetist, Rotkreuzklinikum München gGmbH
Other Study IDs: RotkreuzklinikumMunchen
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Labour Analgesia, Epidural Anaesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women during labour: Women receiving lumbar epidural anaesthesia for pain during birth
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective observational study

SUMMARY:
This is a small observational study investigating the physical changes that occur to epidural catheters after insertion for obstetric anaesthesia. Using the observed physical changes as a correlate for the position of the catheter in the patient we will investigate a connection between the position and e function during labour. This information may be useful in guiding the physicians responses to epidurals that do not provide adequate analgesia to aid in deciding on the most appropriate action

ELIGIBILITY:
Inclusion Criteria:

* any women in labour requesting epidural anaesthesia

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women who request epidural analgesia during birth are eligible
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Position of epidural catheter | directly after removal of the epidural
  the structural form of the epidural catheter will be noted
Analgesia effectiveness | directly after removal of the epidural
  All women will be asked about the effectiveness of the epidural catheter during birth

SECONDARY OUTCOMES:
secondary caesarean section | directly after removal of the epidural
  the proportion of epidurals that were subsequently used for a caesarean section
Impact on motor function | directly after removal of the epidural
  the effect of the epidural catheter on leg strength and the ability of women to ambulate

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Muggleton, MBChB, Principal Investigator — Anaesthetist Rotkreuzklinikum München
Locations (1):
- Frauenklinik Taxisstrasse, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No